CLINICAL TRIAL: NCT02169557
Title: Efficacy and Safety of Fexinidazole in Patients With Stage 1 or Early Stage 2 Human African Trypanosomiasis (HAT) Due to T.b. Gambiense: a Prospective, Multicentre, Open-label Cohort Study, plug-in to the Pivotal Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNDiHATFEX005
Record Dates: First submitted 2014-05-15; First posted 2014-06-23 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Human African Trypanosomiasis (HAT)
MeSH Terms: interventions — fexinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fexinidazole (Experimental)
  Interventions: Drug: Fexinidazole

INTERVENTIONS:
Drug: Fexinidazole

SUMMARY:
The purpose of this study is to demonstrate the treatment success of fexinidazole, at one year follow-up visit, in HAT stage 1 and early stage 2 patients.

DETAILED DESCRIPTION:
Primary Objective

-To demonstrate that the success rate of fexinidazole at one year follow-up in stage 1 and early stage 2 patients is greater than 80%. An 80 % success rate is considered as unacceptable.

Secondary Objectives

* To verify whether the success rate of fexinidazole treatment depends on the stage of the disease (stage 1 versus early stage 2); and, if the difference between the 2 stages is significant, to show that the success rate is greater than 80% and compatible with the historical success rate of NECT in early stage 2 patients and with the historical success rate of pentamidine in stage 1 patients.
* To verify whether the success rate of fexinidazole treatment depends on the number of WBCs in CSF before treatment initiation.
* To assess changes in the success rate over time.
* To evaluate the safety of fexinidazole and determine whether its safety profile is comparable to the historical safety profile of pentamidine.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 15 years old or more
* Male or female
* Ability to ingest at least one complete meal per day (or at least one Plumpy'Nut® sachet)
* Karnofsky index > 50
* Presence of trypanosomes in blood or lymph
* Absence of trypanosomes in CSF
* Permanent address and ability to comply with the follow-up visit schedule
* Patient agreeing to be hospitalized to receive the treatment

Exclusion Criteria:

* Severely malnutrition, defined as BMI < 16.
* Inability to take oral medication.
* Pregnancy or breastfeeding (a urine pregnancy test will be performed in all women of childbearing age within 24 h prior to treatment).
* Clinically relevant medical condition other than HAT that, in the Investigator's opinion, may jeopardize patient safety or interfere with participation in the study, including but not limited to significant liver or cardiovascular disease, documented or suspected active infection (including AIDS), CNS trauma or seizure disorders, coma or altered consciousness.
* Severely deteriorated general condition, e.g. cardiovascular shock, respiratory distress syndrome, or terminal illness.
* Any medical condition (except HAT specific symptoms) hindering communication with the Investigator as required for the completion of this study.
* Any contraindication to imidazole products (known hypersensitivity to imidazoles).
* History of HAT treatment in the past 2 years.
* Patients previously enrolled in the study or having already received fexinidazole.
* Expected follow-up difficulties (migrants, refugees, itinerant vendors, etc.).
* Current alcohol or drug abuse.
* Clinically significant abnormal laboratory value, such as:
* Alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) > 2 times ULN
* Total bilirubin (TBIL) > 1.5 times ULN
* Severe leukopenia (< 2000/mm3)
* Potassium (K+) < 3.5 mmol/L
* Any clinically significant abnormal value (see details in Investigator Manual)
* Pregnancy confirmed by a positive urine pregnancy test obtained within 24 h prior to start of study treatment (see Section 5.8.3 Contraception; p35) QTcF ≥ 450 ms as measured automatically (if the first measurement is abnormal, a second assessment will be done at least 10-20 min later, with the patient in resting position)
* Patients not tested for malaria and/or not treated adequately for this infection
* Patients not treated adequately for soil-transmitted helminthic diseases

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2016-10-09 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Outcome (success or failure) at the test of cure (ToC) visit 12 months after the end of treatment (EOT). | 12 months after end of treatment (day 11)

SECONDARY OUTCOMES:
Success or failure at each visit between the End of treatment and 18 months visit. | End of treatment (day 11) to last follow-up visit (18 months)

OTHER OUTCOMES:
Safety | From signature of informed consent to 18 months Follow up visit
  * Occurrence of any grade AEs (all grades combined) during the observation period.
  * Occurrence of drug-related AEs (Grade ≥ 3 and any grade) during the observation period.
  * Occurrence of any serious adverse events (SAE) from first drug intake to the end of follow up period (M18).

CONTACTS AND LOCATIONS:
Locations (1):
- Kinshasa, Democratic Republic of the Congo

REFERENCES:
- [Derived] Kande Betu Ku Mesu V, Mutombo Kalonji W, Bardonneau C, Valverde Mordt O, Ngolo Tete D, Blesson S, Simon F, Delhomme S, Bernhard S, Mahenzi Mbembo H, Mpia Moke C, Lumeya Vuvu S, Mudji E'kitiak J, Akwaso Masa F, Mukendi Ilunga M, Mpoyi Muamba Nzambi D, Mayala Malu T, Kapongo Tshilumbwa S, Botalema Bolengi F, Nkieri Matsho M, Lumbala C, Scherrer B, Strub-Wourgaft N, Tarral A. Oral fexinidazole for stage 1 or early stage 2 African Trypanosoma brucei gambiense trypanosomiasis: a prospective, multicentre, open-label, cohort study. Lancet Glob Health. 2021 Jul;9(7):e999-e1008. doi: 10.1016/S2214-109X(21)00208-4. PMID 34143998